CLINICAL TRIAL: NCT03642717
Title: A Regulatory Requirement Non Interventional Study to Monitor the Safety and Effectiveness of JARDIANCE DUO® (Empagliflozin/Metformin, 5/500mg, 5/850mg, 5/1000mg, 12.5/500mg, 12.5/850mg, 12.5/1000mg) in Korean Patients With Type 2 Diabetes Mellitus
Brief Title: Regulatory Request NIS in Korea
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1276-0039
Record Dates: First submitted 2018-08-17; First posted 2018-08-22 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects diagnosed with type 2 diabetes mellitus
  Interventions: Drug: JARDIANCE DUO®

INTERVENTIONS:
Drug: JARDIANCE DUO® — empagliflozin and metformin

SUMMARY:
To monitor the safety profile and effectiveness of JARDIANCE DUO® in Korean patients with type 2 diabetes mellitus in a routine clinical practice setting

ELIGIBILITY:
Inclusion Criteria:

* Patients who have started at first time on JARDIANCE DUO® in accordance with the approved label in Korea
* Age ≥19 years at enrolment
* Patients who have signed on the data release consent form

Exclusion Criteria:

* Patients with previous exposure to JARDIANCE®, JARDIANCE DUO®
* Hypersensitivity to active ingredients empagliflozin and/or metformin or to any of the excipients
* Moderate (stage 3b) and severe renal failure (CrCl < 45 ml/min or eGFR < 45 ml/min/1.73 square meter)
* Acute conditions with the potential to alter renal function such as: dehydration, severe infection, cardiovascular collapse (shock), acute myocardial infarction, sepsis
* Type1 diabetes, acute or chronic metabolic acidosis, including diabetic ketoacidosis with or without coma, history of a ketoacidosis (type 1 diabetes and diabetic ketoacidosis should be treated with insulin).
* Congestive heart failure requiring pharmacologic management, in particular those with unstable or acute congestive heart failure
* Radiologic studies involving the use of intravascular iodinated contrast materials (for example, intravenous urogram, intravenous cholangiography, angiography, and computed tomography (CT) scans with intravascular contrast materials)
* Intravascular administration of iodinated contrast media may lead to acute renal failure and has been associated with lactic acidosis in patients receiving metformin.

Therefore, in patients with eGFR > 60ml/min/1.73m2, JARDIANCE DUO® must be discontinued prior to, or at the time of the test and not be reinstituted until 48 hours afterwards, and only after renal function has been re-evaluated and has not deteriorated further. In patients with moderate renal impairment (eGFR 45-60 ml/min/1.73m2), JARDIANCE DUO® must be discontinued 48 hours before administration of iodinated contrast media and not be reinstituted until at least 48 hours afterwards, and only after renal function has been re-evaluated and has not deteriorated further.

* In patients with severe infections or severe traumatic systemic disorders, JARDIANCE DUO® should be temporarily suspended, and should not be restarted until the patient's oral intake has resumed and renal function has been evaluated as normal.
* JARDIANCE DUO® should be temporarily suspended for any surgical procedure(except minor procedures not associated with restricted intake of food and fluids)before 48 hours, and not be reinstituted until 48 hours afterwards, after renal function has been evaluated as normal.
* Patients with malnutrition, starvation, hypostheniam pituitary or adrenal insufficiency
* Impaired hepatic function (since impaired hepatic function has been associated with some cases of lactic acidosis, JARDIANCE DUO® should generally be avoided in patients with clinical or laboratory evidence of hepatic disease), pulmonary infarction, severe respiratory impairment, any condition associated with hypoxemia, excessive alcohol intake, GI disorders such as dehydration, diarrhoea or vomiting
* Pregnant women, women who may be pregnant, nursing women
* Disease which may cause tissue hypoxia (especially acute disease, or worsening of chronic disease) such as: decompensated heart failure, respiratory failure, recent myocardial infarction, shock
* Current participation in other clinical trials

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational prospective, non-interventional, open-label, multi-centre national study. It will provide additional safety information of JARDIANCE DUO® (empagliflozin/metformin) in Korean patients with type 2 diabetes mellitus in a routine clinical practice setting
Sampling Method: Non-Probability Sample
Enrollment: 658 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane(JiEun) Lee, 8227090092, Study Chair — jane.lee.ext@boehringer-ingelheim.com
Locations (20):
- South Korea (20):
  - Korea University Ansan Hospital, Ansan
  - Hyewon Medical Foundation Sejong Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Eulji University Hospital, Daejeon
  - Myongji Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Inje University Sanggye Paik Hospital, Seoul
  - Seoul Medical Center, Seoul
  - Kyung Hee University Hospital, Seoul
  - SoonChunHyang University Seoul Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Hongik Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). Requestors can use the following link http://trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement.

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This post-marketing surveillance study re-examined case report forms retrieving at 20 sites from 21 January 2016 till 11 August 2020 for subjects who had Type 2 Diabetes Mellitus, and were initially administered Jardiance Duo® following the study start date investigating factors affecting the safety and effectiveness of study drug.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- JARDIANCE DUO® (Empagliflozin/Metformin): All subjects who had Type 2 Diabetes Mellitus (T2DM), were initially administered orally various dosages of Jardiance Duo® tablet (Jardiance Duo® (empagliflozin/metformin) tablet dosages: 5/500 milligrams (mg), 5/850 mg, 5/1000 mg, 12.5/500 mg, 12.5/850 mg, 12.5/1000 mg) following the baseline (Visit 1) for an administration for 24 weeks, and with the case report forms (CRFs) retrieving at 20 sites from 21 January 2016 till 11 August 2020. Each patient was planned to be visited once at baseline (Visit 1), followed by 2 planned follow-up visits at Week 12 (after 12 weeks of medication administration) and at Week 24 (after 24 weeks of medication administration).
Period: Overall Study
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Started | 658
Completed | 620
Not Completed | 38
Not completed — Lost to Follow-up | 2
Not completed — Inclusion/exclusion criteria violation | 33
Not completed — Taken study drug prior to contract date | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set: this set included those who signed the informed consent form to participate in this study as subject, took Jardiance Duo® once at least, and were followed up by the physician once or more.
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 620
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.39 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221
  Male | 399
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Adverse Events
Description: Percentage of participants with any adverse events was reported. The 95% Confidence Interval for the percentage of participants with adverse event was calculated by Exact Method.
Time Frame: From baseline (Visit 1) until last visit (the last follow-up visit a patient actually received during the study), up to 349 days.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 620
Percentage of participants | 11.94 [9.49 to 14.75]

2. Primary Outcome: Percentage of Participants With Adverse Events Relating to Study Drug
Description: Percentage of participants with adverse events relating to study drug was reported. The 95% Confidence Interval for the percentage of participants with adverse event was calculated by Exact Method.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- JARDIANCE DUO® (Empagliflozin/Metformin): All subjects who had Type 2 Diabetes Mellitus (T2DM), were initially administered orally various dosages of Jardiance Duo® tablet (Jardiance Duo® (empagliflozin/metformin) tablet dosages: 5/500 milligrams (mg), 5/850 mg, 5/1000 mg, 12.5/500 mg, 12.5/850 mg, 12.5/1000 mg) following the baseline (Visit 1) for an administration for 24 weeks, and with the case report forms (CRFs) retrieving at 20 sites from 21 January 2016 till 11 August 2020. Each patient was visited once at baseline (Visit 1), followed by 1 follow-up visit at 12 weeks after baseline (after 12 weeks of treatment), and the last visit of the study at 24 weeks after baseline (after 24 weeks of treatment).
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 620
Percentage of participants | 5.48 [3.83 to 7.58]

3. Primary Outcome: Percentage of Participants With Unexpected Adverse Events
Description: Percentage of participants with unexpected adverse events was reported. The 95% Confidence Interval for the percentage of participants with adverse event was calculated by Exact Method.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 620
Percentage of participants | 9.03 [6.89 to 11.57]

4. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest
Description: Percentage of participants with adverse events of special interest was reported. The 95% Confidence Interval for the percentage of participants with adverse event was calculated by Exact Method.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 620
Percentage of participants | 0.65 [0.18 to 1.64]

5. Primary Outcome: Percentage of Participants With Adverse Events Leading to Discontinuation of the Drug
Description: Percentage of participants with adverse events leading to discontinuation of the drug was reported. The 95% Confidence Interval for the percentage of participants with adverse event was calculated by Exact Method.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 620
Percentage of participants | 2.90 [1.73 to 4.55]

6. Secondary Outcome: Change in the Glycosylated Hemoglobin (HbA1c) at Last Visit From Baseline
Description: Change in the glycosylated hemoglobin (HbA1c) at Last Visit from baseline was reported.
Time Frame: At baseline (Visit 1) and at last visit (the last follow-up visit a patient actually received during the study, up to Day 349 after baseline).
Population: Effective analysis set: this set included those who signed the informed consent form to participate in this study as subject, took Jardiance Duo®, and were evaluated for the effectiveness.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 497
Percentage of glycosylated hemoglobin | -0.72 (1.47)
Statistical Analysis 1: Comparison: JARDIANCE DUO® (Empagliflozin/Metformin); Test type: Other; p < 0.0001, Paired t-test — Paired t-test was applied comparing the difference in mean of change in Glycosylated hemoglobin (HbA1c) at Last Visit versus at Baseline

7. Secondary Outcome: Number of Participants Reached Target Effectiveness Response in the Glycosylated Hemoglobin (HbA1c) (HbA1c < 7%) at Last Visit
Description: Number of participants reached target effectiveness response in the glycosylated hemoglobin (HbA1c) (HbA1c < 7%) at Last Visit was reported. Target effectiveness response in the glycosylated hemoglobin (HbA1c) was defined as HbA1c less than 7%.
Time Frame: At last visit (the last follow-up visit a patient actually received during the study, up to Day 349 after baseline).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 497
Participants
  less than 7% | 239
  greater than or equal to 7% | 258

8. Secondary Outcome: Number of Participants With Relative Effectiveness Response in the Glycosylated Hemoglobin (HbA1c) (HbA1c Decrease of 0.5% Comparing to Baseline) at Last Visit
Description: Number of participants with relative effectiveness response in the glycosylated hemoglobin (HbA1c) at Last Visit was reported. Relative effectiveness response in the glycosylated hemoglobin (HbA1c) at last visit was defined as HbA1c decrease of 0.5% or more at the last visit comparing to baseline.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 497
Participants
  greater than or equal to 0.5% | 242
  less than 0.5% | 255

9. Secondary Outcome: Change in the Fasting Plasma Glucose (FPG) at Last Visit From Baseline
Description: Change in the Fasting Plasma Glucose (FPG) at Last Visit from baseline was reported.
Time Frame: as for outcome 6
Population: Effective analysis set: this set included those who signed the informed consent form to participate in this study as subject, took Jardiance Duo®, and were evaluated for the effectiveness. Only those subjects with non-missing outcome measures were included in this analysis.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dl)
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 417
milligrams per deciliter (mg/dl) | -26.86 (50.91)
Statistical Analysis 1: Comparison: JARDIANCE DUO® (Empagliflozin/Metformin); Test type: Other; p < 0.0001, Paired t-test — Paired t-test was applied comparing the difference in mean of change in Fasting Plasma Glucose (FPG) at Last Visit versus at Baseline

10. Secondary Outcome: Change in the Body Weight at Last Visit From Baseline
Description: Change in the body weight at Last Visit from baseline was reported.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 372
kilogram (kg) | -2.18 (3.53)
Statistical Analysis 1: Comparison: JARDIANCE DUO® (Empagliflozin/Metformin); Test type: Other; p < 0.0001, Paired t-test — Paired t-test was applied comparing the difference in mean of change in body weight at Last Visit versus at Baseline

11. Secondary Outcome: Change in the Systolic Blood Pressure (SBP) at Last Visit From Baseline
Description: Change in the systolic blood pressure (SBP) at Last Visit from baseline was reported.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 448
millimetre of mercury (mmHg) | -1.96 (15.45)
Statistical Analysis 1: Comparison: JARDIANCE DUO® (Empagliflozin/Metformin); Test type: Other; p = 0.0076, Paired t-test — Paired t-test was applied comparing the difference in mean of change in systolic blood pressure (SBP) at Last Visit versus at Baseline

12. Secondary Outcome: Change in the Diastolic Blood Pressure (DBP) at Last Visit From Baseline
Description: Change in the diastolic blood pressure (DBP) at Last Visit from baseline was reported.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 448
millimetre of mercury (mmHg) | -2.04 (10.80)
Statistical Analysis 1: Comparison: JARDIANCE DUO® (Empagliflozin/Metformin); Test type: Other; p < 0.0001, Paired t-test — Paired t-test was applied comparing the difference in mean of change in diastolic blood pressure (DBP) at Last Visit versus at Baseline

13. Secondary Outcome: Number of Participants Per Final Effectiveness Assessment Category at Last Visit
Description: Number of participants per final effectiveness assessment category at Last Visit was reported. The final effectiveness consisted of 4 categories: Improved (If determined as there was any effect of maintaining or improving disease related factors.), Unchanged (If disease related factors had not been changed compared with before administration, and not determined as there was any effect of maintaining symptoms.), Aggravated (If disease related factors were worse than before administration.), and Unassessable (If it cannot be determined due to insufficient information collected.).
Time Frame: At last visit (the last follow-up visit a patient actually received during the study, up to Day 349 after baseline).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
Number analyzed (Participants) | 497
Participants
  Improved | 330
  Unchanged | 103
  Aggravated | 45
  Unassessable | 19

ADVERSE EVENTS:
Time Frame: From baseline (Visit 1) until last visit (the last follow-up visit a patient actually received during the study), up to 349 days.
Description: Safety analysis set: this set included those who signed the informed consent form to participate in this study as subject, took Jardiance Duo® once at least, and were followed up by the physician once or more.
Arm/Group | JARDIANCE DUO® (Empagliflozin/Metformin)
All-Cause Mortality (participants affected / at risk) | 0/620
Serious Adverse Events (participants affected / at risk) | 10/620
Other Adverse Events (participants affected / at risk) | 0/620
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JARDIANCE DUO® (Empagliflozin/Metformin) (N=620)
Myocardial infarction (Cardiac disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT03642717/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03642717/SAP_001.pdf